CLINICAL TRIAL: NCT05152199
Title: The Assessment of Pain Outcomes During Rigid Cystoscopy in Females With and Without the Use of the Rigid Cystoscope Obturator: A Randomized Control Trial
Brief Title: Pain Outcomes During Rigid Cystoscopy in Females With and Without Cystoscopic Sheath Obturator
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI employment status change inhibiting continued recruitment
Sponsor: Todd Moyerbrailean DO FACOG (Other)
Responsible Party: Sponsor-Investigator, Todd Moyerbrailean DO FACOG, Associate Professor, Michigan State University
Organization: Michigan State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00005662
Record Dates: First submitted 2021-11-23; First posted 2021-12-09 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Dysuria
Keywords: Rigid Cystoscopy; Obturator Sheath; Urogynecology
MeSH Terms: conditions — Dysuria | interventions — Cystoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cystoscopy with use of obturator sheath (Other): This intervention arm will include the use of the obturator sheath upon entry into the urethra during rigid cystoscopy.
  Interventions: Procedure: Cystoscopy - with use of obturator sheath
- Cystoscopy without use of obturator sheath (Active Comparator): This intervention arm will not include the use of the obturator sheath upon entry into the urethra during rigid cystoscopy, but will consist of using the telescope under direct visualization.
  Interventions: Procedure: Cystoscopy - without use of obturator sheath

INTERVENTIONS:
Procedure: Cystoscopy - with use of obturator sheath — The intervention arm will include the use of the obturator sheath upon entry into the urethra during rigid cystoscopy.
  Arms: Cystoscopy with use of obturator sheath
Procedure: Cystoscopy - without use of obturator sheath — The intervention arm will not include the use of the obturator sheath upon entry into the urethra during rigid cystoscopy, but will consist of using the telescope under direct visualization.
  Arms: Cystoscopy without use of obturator sheath

SUMMARY:
Rigid cystoscopy is a common procedure to evaluate lower urinary tract symptoms in females. This procedure can be done with or without an instrument called a sheath obturator. Both techniques are used by surgeons and are considered safe, but have never been studied to see if one technique leads to less discomfort with the patient's first void after the procedure. The obturator's use may potentially reduce urethral irritation and bothersome postprocedural symptoms, primarily dysuria. The investigators aim to determine whether there is a difference in dysuria outcomes postoperatively when cystoscopy is performed with or without an obturator.

DETAILED DESCRIPTION:
Rigid cystoscopy is a common procedure to evaluate lower urinary tract symptoms in females. This procedure can be done with or without an instrument called a sheath obturator (or obturator for short). There are two acceptable insertion techniques for performing cystoscopy in women. Surgeons can perform cystoscope without the use of the obturator by using a "visual" technique where a telescope with a sheath is inserted for entry into the bladder (referred to as cystoscopy without the obturator). Surgeons can also perform cystoscopy by using an obturator with a sheath allowing for smooth entry without needing the telescope (referred to as cystoscopy with the obturator). Both techniques are used by surgeons and are considered safe, but have never been studied to see if one technique leads to less discomfort with the patient's first void after the procedure. The obturator's use may potentially reduce urethral irritation and bothersome postprocedural symptoms, primarily dysuria. The investigators aim to determine whether there is a difference in dysuria outcomes postoperatively when cystoscopy is performed with or without an obturator.

ELIGIBILITY:
Inclusion Criteria:

* Female patients scheduled for gynecological procedures where cystoscopy is indicated
* Ability to comprehend and participate in the study

Exclusion Criteria:

* < 18 years
* Pregnancy
* Current pelvic mesh erosion
* Exposure or pain complications from mesh
* Genitourinary malignancy;
* History of recurrent urinary tract infection (e.g., 2 in 6 months)

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Post-Procedure Dysuria | Post intervention pain scale assessment within 10 minutes following first void after the procedure.
  The participant will be asked to void within 10 minutes of the completed procedure. The participant will then complete a Visual Analog Numeric Pain Scale, where 1 = no pain and 10 = worst possible pain, within 10 minutes of voiding.

SECONDARY OUTCOMES:
Strength of stream | Within 10 minutes following the first post-procedure void.
  A 6 item questionnaire will be completed within 10 minutes following the first post-procedure void and include a multiple choice question assessing the participants strength of stream as: 1 - not reduced, 2 - reduced a little, 3 - quite reduced, 4 - reduced a great deal, 5 - I had no stream
Bladder pain | Within 10 minutes following the first post-procedure void.
  A 6 item questionnaire will be completed within 10 minutes following the first post-procedure void and include a yes/no question "Do you have pain in your bladder?"
Hesitancy | Within 10 minutes following the first post-procedure void.
  A 6 item questionnaire will be completed within 10 minutes following the first post-procedure void and include a yes/no question "Was there a delay before you started to urinate?"
Straining | Within 10 minutes following the first post-procedure void.
  A 6 item questionnaire will be completed within 10 minutes following the first post-procedure void and include a yes/no question "Did you have to strain to start urinating?"
Incomplete Emptying | Within 10 minutes following the first post-procedure void.
  A 6 item questionnaire will be completed within 10 minutes following the first post-procedure void and include a yes/no question "Did you feel that your bladder was empty after urinating?"
Post-procedure pain | Within 10 minutes following completion of the procedure
  The participant will be asked to complete a Visual Analog Numeric Pain Scale, where 1 = no pain and 10 = worst possible pain, within 10 minutes of procedure completion.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Moyerbrailean, DO, FACOG, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be shared with members of the investigation team.

REFERENCES:
- [Background] Ellerkmann RM, Dunn JS, McBride AW, Kummer LG, Melick CF, Bent AE, Blomquist JL. A comparison of anticipated pain before and pain rating after the procedure in patients who undergo cystourethroscopy. Am J Obstet Gynecol. 2003 Jul;189(1):66-9. doi: 10.1067/mob.2003.377. PMID 12861140
- [Background] Nguyen CT, Babineau DC, Jones JS. Impact of urologic resident training on patient pain and morbidity associated with office-based cystoscopy. Urology. 2008 May;71(5):782-6. doi: 10.1016/j.urology.2007.12.032. PMID 18455622
- [Background] Quiroz LH, Shobeiri SA, Nihira MA, Brady J, Wild RA. Randomized trial comparing office flexible to rigid cystoscopy in women. Int Urogynecol J. 2012 Nov;23(11):1625-30. doi: 10.1007/s00192-012-1777-0. Epub 2012 May 9. PMID 22569690
- [Background] Yerlikaya G, Laml T, Elenskaia K, Hanzal E, Kolbl H, Umek W. Pain perception during outpatient cystoscopy: a prospective controlled study. Eur J Obstet Gynecol Reprod Biol. 2014 Feb;173:101-5. doi: 10.1016/j.ejogrb.2013.11.007. Epub 2013 Nov 14. PMID 24300559
- [Background] Greenstein A, Greenstein I, Senderovich S, Mabjeesh NJ. Is diagnostic cystoscopy painful? Analysis of 1,320 consecutive procedures. Int Braz J Urol. 2014 Jul-Aug;40(4):533-8. doi: 10.1590/S1677-5538.IBJU.2014.04.13. PMID 25251958
- [Background] Seklehner S, Remzi M, Fajkovic H, Saratlija-Novakovic Z, Skopek M, Resch I, Duvnjak M, Hruby S, Librenjak D, Hubner W, Breinl E, Riedl C, Engelhardt PF. Prospective multi-institutional study analyzing pain perception of flexible and rigid cystoscopy in men. Urology. 2015 Apr;85(4):737-41. doi: 10.1016/j.urology.2015.01.007. PMID 25817101
- [Background] Casteleijn NF, Vriesema JL, Stomps SP, van Balen OL, Cornel EB. The effect of office based flexible and rigid cystoscopy on pain experience in female patients. Investig Clin Urol. 2017 Jan;58(1):48-53. doi: 10.4111/icu.2017.58.1.48. Epub 2017 Jan 4. PMID 28097268
- [Background] Dougher E, Zoorob D, Thomas D, Hagan J, Peacock L. The Effect of Lidocaine Gel on Pain Perception During Diagnostic Flexible Cystoscopy in Women: A Randomized Control Trial. Female Pelvic Med Reconstr Surg. 2019 Mar/Apr;25(2):178-184. doi: 10.1097/SPV.0000000000000680. PMID 30807424
- [Background] Rappaport YH, Beberashvili I, Zisman A, Stav K. Is Meatal Analgesia Necessary for Pain Reduction During Cystoscopy in Females? A Prospective Randomized Study. Urology. 2020 Dec;146:79-82. doi: 10.1016/j.urology.2020.08.052. Epub 2020 Sep 11. PMID 32920032